CLINICAL TRIAL: NCT05689970
Title: LESTONNAC Study: Observed ST Elevation Does Not Require Acute Cardiac Necrosis
Brief Title: ST-segment Elevation Not Associated With Acute Cardiac Necrosis (LESTONNAC)
Acronym: LESTONNAC
Status: Active, not recruiting | Type: Observational
Sponsor: Idoven 1903 S.L. (Industry)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); Spanish Society of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: 350/21
Record Dates: First submitted 2022-12-20; First posted 2023-01-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: ST segment elevation; Artificial intelligence; Electrocardiogram; Acute myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STE patients: Patients with ST segment elevation (STE) and coronary arteries without significant lesions and without a serum troponin curve suggestive of acute necrosis (group without acute myocardial necrosis).
  Interventions: Diagnostic Test: AI platform to detect ST elevation in ECG
- STEMI patients: Patients with ST segment elevation with acute occlusion of at least one epicardial coronary artery and TIMI flow 0 or I (group with acute myocardial necrosis of ischemic origin), that meet the definition of myocardial infarction (STEMI) with an acute cardiac necrosis curve verified by measurement of troponin I or troponin T.
  Interventions: Diagnostic Test: AI platform to detect ST elevation in ECG

INTERVENTIONS:
Diagnostic Test: AI platform to detect ST elevation in ECG — A clinical decision support software as a medical device that detects whether a patient has ST elevation due to acute myocardial ischemia or due to another etiology based upon the input of one or more ECGs and other clinical data obtained at the point-of-care.
  Other Names: Willem platform; Idoven AI

SUMMARY:
Patients with chest pain and persistent ST segment elevation (STE) may not have acute coronary occlusions or serum troponin curves suggestive of acute necrosis. Our objective is the validation and cost-effectiveness analysis of a diagnostic model assisted by artificial intelligence (AI). Our hypothesis is that an AI analysis of the surface electrocardiogram allows a better distinction of patients with STE due to acute myocardial ischemia, from those with another etiology. This is a prospective multicenter study with two groups of patients with STE: I) coronary arteries without significant lesions and without serum troponin curve suggestive of acute necrosis, II) myocardial infarction with acute coronary occlusion. A manual centralized electrocardiographic analysis and another by AI algorithms will be performed.

DETAILED DESCRIPTION:
This is a prospective multicenter study promoted by the Ischemic Heart Disease and Acute Cardiovascular Care Section of the Spanish Society of Cardiology. Following institutional ethical approval, the surface ECG prior to the activation of the Infarction Code, and the ECGs before and after (up to a maximum of 20) the Infarction Code along with other clinical data will be collected across the different enrolled hospitals. Sites will securely transfer the data to a centralized repository for processing. Willem AI platform will automatically analyze the ECGs in parallel to an experienced observer. The results of the study will provide new information for the improvement in the stratification of patients with ST segment elevation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years.
* Chest pain or symptoms suggestive of myocardial ischemia.
* STE at point J in the12-lead electrocardiogram prior to activation of the infarction code in two contiguous leads ≥0.1 mV, in V2 and V3 ≥0.2 mV.
* Signature of informed consent.

Exclusion Criteria:

* Left bundle branch block.
* Acute cardiac necrosis in the absence of significant epicardial coronary artery stenosis >70% (vasospasm, takotsubo stress cardiomyopathy, myocarditis, coronary artery dissection, acute myocardial infarction without obstructive coronary lesions - MINOCA).
* STE≤0.1 mV with pathologic Q wave suggestive of previous chronic infarction.
* Severe anemia (hemoglobin <8.0 g/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients going to the hospital with suspected symptoms of myocardial infarction and ST segment elevation in the electrocardiogram.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-07-24 (Estimated)

PRIMARY OUTCOMES:
Clinical validation of a screening model assisted by AI | 6 months after the last enrolled patient
  The detection performance of acute myocardial ischemia will be evaluated for the AI platform in comparison to standard manual analysis.

SECONDARY OUTCOMES:
Cost-effectiveness analysis of a screening model assisted by AI | 1 year after the last enrolled patient
  The benefits of the screening model assisted by the AI platform will be evaluated using a hybrid decision tree/ Markov model.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Martínez-Sellés, MD, Principal Investigator — Hospital Universitario Gregorio Marañón
Locations (7):
- Spain (7):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Vall D' Hebron, Barcelona
  - Idoven, Madrid
  - Servicio Cardiología Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Selles M, Bueno H, Sacristan A, Estevez A, Ortiz J, Gallego L, Fernandez-Aviles F. Chest pain in the emergency department: incidence, clinical characteristics and risk stratification. Rev Esp Cardiol. 2008 Sep;61(9):953-9. English, Spanish. PMID 18775237
- [Background] Lillo-Castellano JM, Gonzalez-Ferrer JJ, Marina-Breysse M, Martinez-Ferrer JB, Perez-Alvarez L, Alzueta J, Martinez JG, Rodriguez A, Rodriguez-Perez JC, Anguera I, Vinolas X, Garcia-Alberola A, Quintanilla JG, Alfonso-Almazan JM, Garcia J, Borrego L, Canadas-Godoy V, Perez-Castellano N, Perez-Villacastin J, Jimenez-Diaz J, Jalife J, Filgueiras-Rama D. Personalized monitoring of electrical remodelling during atrial fibrillation progression via remote transmissions from implantable devices. Europace. 2020 May 1;22(5):704-715. doi: 10.1093/europace/euz331. PMID 31840163
- [Background] Quartieri F, Marina-Breysse M, Pollastrelli A, Paini I, Lizcano C, Lillo-Castellano JM, Grammatico A. Artificial intelligence augments detection accuracy of cardiac insertable cardiac monitors: Results from a pilot prospective observational study. Cardiovasc Digit Health J. 2022 Aug 4;3(5):201-211. doi: 10.1016/j.cvdhj.2022.07.071. eCollection 2022 Oct. PMID 36310681
- Available data/document: Study Protocol: PubMed ID: 34763217 — https://pubmed.ncbi.nlm.nih.gov/34763217/